CLINICAL TRIAL: NCT02707900
Title: IGHID 11424 - A Pilot Trial of the Effect of Vorinostat and AGS-004 on Persistent HIV-1 Infection (The VOR VAX Study)
Brief Title: Pilot Trial of the Effect of Vorinostat and AGS-004 on Persistent HIV-1 Infection
Acronym: VORVAX
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturing of the AGS-004 HIV vaccine by Argos could no longer be provided.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1626; U01AI117844-01 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-07

CONDITIONS: HIV-1 Infection
Keywords: Vorinostat; AGS-004; HIV virus; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat + AGS-004 (Experimental): Vorinostat (VOR) 400 mg PO - two paired doses at Step 2 (Enrollment) - Only participants demonstrating an in vivo response to the 2nd of the paired VOR doses will proceed to the AGS-004 manufacturing and treatment in Steps 3 through 7.
  Step 4 - AGS-004 vaccination. AGS-004 product will be delivered in three intradermal (ID) injections of 0.2 mL (0.6 mL total volume) for a total of 1.2 x 10-7 viable cells. AGS-004 will be administered every 3 weeks for 4 doses.
  Interventions: Drug: Vorinostat; Biological: AGS-004

INTERVENTIONS:
Drug: Vorinostat — At Step 2 (Enrollment) - subjects receive two paired oral doses of Vorinostat (VOR) 400 mg.
  Step 5 - Approximately 7- 10 days after the 4th dose of AGS-004 in Step 4 (Visit 11), ten (10) doses of VOR 400 mg will be administered at 72 hour intervals.
  Steps 6 - 7 & EOS visit - Repeat cycles of AGS-004 and VOR. Participants will undergo a second series of 4 AGS-004 vaccinations (Step 6) followed by 10 doses of VOR 400 mg PO (Step 7).
  Other Names: Zolinza
Biological: AGS-004 — Step 4 - AGS-004 vaccination. AGS-004 product will be delivered in three intradermal injections of 0.2 mL (0.6 mL total volume) for a total of 1.2 x 10-7 viable cells. AGS-004 will be administered every 3 weeks for 4 doses.
  Steps 6 - 7 & EOS visit - Repeat cycles of AGS-004 and VOR. Participants will undergo a second series of 4 AGS-004 vaccinations (Step 6) followed by 10 doses of VOR 400 mg PO (Step 7).

SUMMARY:
The purpose of this research study is to 1) evaluate the safety of a series of injections with the AGS-004 product in combination with a series of Vorinostat doses and 2) to help scientists evaluate ways of reactivating latent (non-acting) HIV virus and determine if the immune system can be made stronger to eliminate the activated HIV virus.

DETAILED DESCRIPTION:
Purpose: Phase I study to measure the potential of AGS-004 combined with Vorinostat to: 1) stimulate expression of persistent proviral HIV from resting CD4+ cells, 2) generate an HIV-specific immune response, and 3) when combined, clear persistent infection in HIV-infected participants in whom viral replication and spread is inhibited by uninterrupted antiretroviral therapy (ART).

This is a phase I, single-site, pilot study intended to evaluate the association of serial AGS-004 vaccinations in combination with serial VOR doses on the expression of persistent proviral HIV, HIV-specific immune responses, and the frequency of resting CD4+T cell infection. Twelve participants with durable viral suppression will be enrolled. All participants will receive the same treatment and doses of AGS-004 and VOR and continue their baseline ART regimen throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of HIV-1 infection HIV infection is defined as documentation by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

   NOTE: The term "licensed" refers to a US FDA-approved kit.

   WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (eg, indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
2. Ages ≥ 18 to < 65 years old.
3. Karnofsky performance status >70.
4. Ability and willingness of participant to give written informed consent. Note: Due to the lack of foreseeable benefit to study volunteers, illiterate or mentally incompetent volunteers will not be enrolled.
5. Able and willing to provide adequate locator information.
6. On antiretroviral therapy (ART) for at least 24 months and on potent ART for > or equal to 6 months prior to Screening (Visit 1).

   Note: Potent ART is defined by current treatment guidelines and consists of at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor without interruption (defined as missing doses for more than two (2) consecutive days or more than four (4) cumulative days) in the 24 weeks immediately prior to Screening (Visit 1). Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, toxicity, or other reasons are permitted if an alternative suppressive regimen was maintained.
7. All participants must continue cART throughout the study.
8. Able and willing to adhere to protocol therapy and judged adherent to antiretroviral therapy.
9. Plasma HIV-1 RNA < 50 copies/mL at screening (Visit 1).
10. Plasma HIV-1 RNA< 50 copies/mL at two time points in the previous 12 months prior to study screening and never > or equal to 50 copies/mL on two consecutive time points in the last 24 months prior to screening.

    Note: A single unconfirmed plasma HIV RNA > or equal to 50 copies (c)/mL but < 1000 c/mL is allowed if a subsequent assay was < 50 c/mL but not in the 6 months preceding the study screening visit (Visit 1).
11. CD4+ cell count ≥ 300 cells/mm3 at screening (Visit 1).
12. No history of auto-immune disease or auto-immune manifestations.
13. No active HCV infection (HCV antibody negative or no measureable HCV RNA) at or within 90 days of screening (Visit 1).
14. No active HBV infection (measureable HBV DNA or HBVsAg+) at or within 90 days of screening (Visit 1).
15. Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.
16. Adequate vascular access for leukapheresis.
17. Able to swallow pills without difficulty.
18. Able and willing to receive Intradermal (ID) injections without difficulty.
19. Women with written documentation of any of the following:

    1. prior hysterectomy OR bilateral oophorectomy (removal of both ovaries)
    2. bilateral tubal ligation or non-surgical permanent sterilization
    3. Women with intact uterus and ovaries who have not had a period for ≥ one year AND have a documented FSH level indicating postmenopausal status.
20. All male study volunteers must agree not to participate in a conception process (e.g. active attempt to impregnate, sperm donation, in vitro fertilization) and, if participating in sexual activity that could lead to pregnancy, the male study volunteer and his female partner must use two reliable methods of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; or hormonal-based contraception) simultaneously while receiving the protocol-specified study products and for 6 weeks after stopping the study products. Participants must use a reliable barrier method of contraception (condom, cervical cap) along with another form of contraception.

    For the female partners of male study volunteers who are receiving ritonavir, estrogen-based contraceptives are not reliable and an alternative method should be suggested.
21. Potential participant must have adequate organ function as indicated by the following laboratory values:

System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥125,000 / mcL Hemoglobin ≥ 12 g/dL (males) and ≥ 11.5 g/dL (females) Coagulation Prothrombin Time or INR ≤1.1 x upper limit of normal (ULN) Chemistry K+ levels Within normal limits Mg++ levels ≥ 1.4 mEq/L Glucose Screening serum glucose ≤ Grade 1 (fasting or non-fasting) Albumin ≥ 3.5 g/dL Renal Creatinine clearance determined eGFR > 60mL/min by the CKD-Epi equation found at: https://www.qxmd.com/calculate/calculator_ 251/egfr-using-ckd-epi Hepatic Serum total bilirubin Total bilirubin <1.1 X ULN range, unless history of Gilbert's disease or deemed related to treatment with atazanavir. If total bilirubin is elevated, direct bilirubin must be <2 X ULN range.

AST (SGOT) and ALT (SGPT) <1.25 X ULN Lipase <1.1 X ULN Alkaline Phosphatase <1.25 X ULN

Exclusion Criteria:

1. Known allergy or sensitivity to the components of the investigational immunotherapy or the components of VOR or its analogs or DMSO.
2. HIV-2 antibody positive in the absence of a positive HIV-1 Western Blot as measured at the Screening Visit (Visit 1).
3. Untreated syphilis infection (defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment).

   Note: In cases of untreated syphilis, participant may re-screen following documentation of adequate treatment of syphilis
4. Received any infusion blood product, immune globulin, or hematopoetic growth factors within 90 days prior to study entry.
5. All women unless there is written documentation of menopause (absence of a period for ≥ one year and FSH level indicating menopause), hysterectomy, oophorectomy, or tubal ligation.
6. All male participants expecting to father children within the projected duration of the study.
7. Use of any of the following within 90 days prior to screening: immunomodulatory, cytokine, or growth stimulating factors such as systemic cytotoxic chemotherapy, systemic corticosteroids, immune globulin, interferon, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, IFN, interleukins, interleukin-2 (IL-2), hydroxyurea, thalidomide, sargramostim (granulocyte macrophage-colony stimulating factor [GM-CSF]), growth factors, dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin, inosiplex, polyribonucleotide, or ditiocarb sodium, coumadin, warfarin, or other Coumadin derivative anticoagulants.
8. Use of the following medications that carry risk of torsade des pointes: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainimide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.
9. Receipt of compounds with HDAC inhibitor-like activity, such as valproic acid within 30 days prior to screening. Potential participants may enroll after a 30-day washout period.
10. Use of any investigational antiretroviral agents within 30 days prior to Screening (Visit 1).
11. Use of antiretroviral medications that cannot be co-administered with Vorinostat within the 4 weeks of the first dose and anytime thereafter while on the study.
12. If the HIV care provider or study investigator is unable, as assessed by the study PI or protocol team, to construct a fully active alternative ART regimen based on previous resistance testing and/or treatment history.
13. Use of systemic corticosteroids or use of topical steroids over a total area exceeding 15 cm2 within 30 days prior to Screening, or anticipated need for periodic use of corticosteroids during the study.

    NOTE: For participants receiving ritonavir (as a booster or protease inhibitor (PI) as part of their ART regimen, the concomitant use of oral/systemic/topical/inhaled/intranasal corticosteroids is prohibited.
14. Any serious illness requiring systemic treatment or hospitalization, the participant must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to entry.
15. Known history of a bone marrow disorder
16. Treatment for an active AIDS-defining opportunistic infection within 90 days prior to Screening.
17. Any active malignancy that may require chemotherapy or radiation therapy.
18. History of lymph node irradiation or dissection.
19. Evidence of hepatic decompensation in cirrhotic participants: history of ascites, hepatic encephalopathy, or bleeding esophageal varices.
20. History or other clinical evidence of significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia) or clinically significant electrocardiogram (ECG) abnormalities. Any history of cardiac rhythm disturbance requiring medical or surgical therapy.
21. Any history of acute or chronic pancreatitis.
22. Any renal disorder deemed clinically significant by the investigator.
23. Active autoimmune disease or condition including, but not limited to:

    Rheumatoid arthritis (RF positive arthritis with current or recent flare); Inflammatory bowel disease/ulcerative colitis/Crohn's Disease; Systemic lupus erythematosis (clinical evidence confirmed with ANA >1:80); Ankylosing spondylitis; Hashimoto's disease; Scleroderma; Multiple sclerosis; Autoimmune hemolytic anemia (AHA); Thyroiditis Immune thrombocytopenic purpura; and, Type I diabetes mellitus (insulin therapy for Type II diabetes is permitted).
24. History or other evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the participant unsuitable for the study in the opinion of the investigator (or designee) Note: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary with documentation of complete resection.
25. History of neoplastic disease with extensive involvement of the bone marrow or lymphatic system or participants severely compromised hematopoietic function.
26. Inability to communicate with study personnel.
27. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease.
28. Prisoner recruitment and participation is not permitted.
29. Known psychiatric or substance abuse disorders that would interfere with participant's ability to fully cooperate with the requirements of the trial as assessed by the study investigator (or designee).
30. Participation in another investigational clinical research study (with the exception of an antiretroviral treatment trial that uses FDA approved antiretroviral agents) or use of investigational agents within 30 days prior to Screening (Visit 1).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of HIV infection per million resting CD4+T cells (RCI) from baseline to post-VOR/AGS. | First day of study treatment to between approximately week 43 and week 72 on study
  Change in the frequency of HIV infection per million resting CD4+T cells (RCI) from baseline to post-VOR/AGS.
Occurrence of at least one ≥ Grade 3 adverse event including signs/symptoms, lab toxicities, and/or clinical events that is possibly or definitely related to VOR or AGS-004 any time from the first day of study treatment through the end of study. | First day of study treatment to between approximately week 73 and week 96 on study
  Safety data will include local and systemic signs and symptoms, laboratory measures of safety/toxicity, and all adverse and serious adverse events. Safety data will be routinely collected throughout the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David M Margolis, MD, FACP, Principal Investigator — University of North Carolina, Chapel Hill; Cynthia L Gay, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Finzi D, Blankson J, Siliciano JD, Margolick JB, Chadwick K, Pierson T, Smith K, Lisziewicz J, Lori F, Flexner C, Quinn TC, Chaisson RE, Rosenberg E, Walker B, Gange S, Gallant J, Siliciano RF. Latent infection of CD4+ T cells provides a mechanism for lifelong persistence of HIV-1, even in patients on effective combination therapy. Nat Med. 1999 May;5(5):512-7. doi: 10.1038/8394. PMID 10229227
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Gay CL, DeBenedette MA, Tcherepanova IY, Gamble A, Lewis WE, Cope AB, Kuruc JD, McGee KS, Kearney MF, Coffin JM, Archin NM, Hicks CB, Eron JJ, Nicolette CA, Margolis DM. Immunogenicity of AGS-004 Dendritic Cell Therapy in Patients Treated During Acute HIV Infection. AIDS Res Hum Retroviruses. 2018 Jan;34(1):111-122. doi: 10.1089/aid.2017.0071. Epub 2017 Jun 21. PMID 28636433
- [Background] Coull JJ, Romerio F, Sun JM, Volker JL, Galvin KM, Davie JR, Shi Y, Hansen U, Margolis DM. The human factors YY1 and LSF repress the human immunodeficiency virus type 1 long terminal repeat via recruitment of histone deacetylase 1. J Virol. 2000 Aug;74(15):6790-9. doi: 10.1128/jvi.74.15.6790-6799.2000. PMID 10888618
- [Background] Romerio F, Gabriel MN, Margolis DM. Repression of human immunodeficiency virus type 1 through the novel cooperation of human factors YY1 and LSF. J Virol. 1997 Dec;71(12):9375-82. doi: 10.1128/JVI.71.12.9375-9382.1997. PMID 9371597
- [Background] He G, Margolis DM. Counterregulation of chromatin deacetylation and histone deacetylase occupancy at the integrated promoter of human immunodeficiency virus type 1 (HIV-1) by the HIV-1 repressor YY1 and HIV-1 activator Tat. Mol Cell Biol. 2002 May;22(9):2965-73. doi: 10.1128/MCB.22.9.2965-2973.2002. PMID 11940654
- [Background] Coull JJ, He G, Melander C, Rucker VC, Dervan PB, Margolis DM. Targeted derepression of the human immunodeficiency virus type 1 long terminal repeat by pyrrole-imidazole polyamides. J Virol. 2002 Dec;76(23):12349-54. doi: 10.1128/jvi.76.23.12349-12354.2002. PMID 12414976
- [Background] Ylisastigui L, Coull JJ, Rucker VC, Melander C, Bosch RJ, Brodie SJ, Corey L, Sodora DL, Dervan PB, Margolis DM. Polyamides reveal a role for repression in latency within resting T cells of HIV-infected donors. J Infect Dis. 2004 Oct 15;190(8):1429-37. doi: 10.1086/423822. Epub 2004 Sep 15. PMID 15378435
- [Background] Ylisastigui L, Archin NM, Lehrman G, Bosch RJ, Margolis DM. Coaxing HIV-1 from resting CD4 T cells: histone deacetylase inhibition allows latent viral expression. AIDS. 2004 May 21;18(8):1101-8. doi: 10.1097/00002030-200405210-00003. PMID 15166525
- [Background] Marban C, Suzanne S, Dequiedt F, de Walque S, Redel L, Van Lint C, Aunis D, Rohr O. Recruitment of chromatin-modifying enzymes by CTIP2 promotes HIV-1 transcriptional silencing. EMBO J. 2007 Jan 24;26(2):412-23. doi: 10.1038/sj.emboj.7601516. PMID 17245431
- [Background] Williams SA, Chen LF, Kwon H, Ruiz-Jarabo CM, Verdin E, Greene WC. NF-kappaB p50 promotes HIV latency through HDAC recruitment and repression of transcriptional initiation. EMBO J. 2006 Jan 11;25(1):139-49. doi: 10.1038/sj.emboj.7600900. Epub 2005 Dec 1. PMID 16319923
- [Background] Imai K, Okamoto T. Transcriptional repression of human immunodeficiency virus type 1 by AP-4. J Biol Chem. 2006 May 5;281(18):12495-505. doi: 10.1074/jbc.M511773200. Epub 2006 Mar 15. PMID 16540471
- [Background] Jiang G, Espeseth A, Hazuda DJ, Margolis DM. c-Myc and Sp1 contribute to proviral latency by recruiting histone deacetylase 1 to the human immunodeficiency virus type 1 promoter. J Virol. 2007 Oct;81(20):10914-23. doi: 10.1128/JVI.01208-07. Epub 2007 Aug 1. PMID 17670825
- [Background] du Chene I, Basyuk E, Lin YL, Triboulet R, Knezevich A, Chable-Bessia C, Mettling C, Baillat V, Reynes J, Corbeau P, Bertrand E, Marcello A, Emiliani S, Kiernan R, Benkirane M. Suv39H1 and HP1gamma are responsible for chromatin-mediated HIV-1 transcriptional silencing and post-integration latency. EMBO J. 2007 Jan 24;26(2):424-35. doi: 10.1038/sj.emboj.7601517. PMID 17245432
- [Background] Tyagi M, Karn J. CBF-1 promotes transcriptional silencing during the establishment of HIV-1 latency. EMBO J. 2007 Dec 12;26(24):4985-95. doi: 10.1038/sj.emboj.7601928. Epub 2007 Nov 15. PMID 18007589
- [Background] Lehrman G, Hogue IB, Palmer S, Jennings C, Spina CA, Wiegand A, Landay AL, Coombs RW, Richman DD, Mellors JW, Coffin JM, Bosch RJ, Margolis DM. Depletion of latent HIV-1 infection in vivo: a proof-of-concept study. Lancet. 2005 Aug 13-19;366(9485):549-55. doi: 10.1016/S0140-6736(05)67098-5. PMID 16099290
- [Background] Siliciano JD, Lai J, Callender M, Pitt E, Zhang H, Margolick JB, Gallant JE, Cofrancesco J Jr, Moore RD, Gange SJ, Siliciano RF. Stability of the latent reservoir for HIV-1 in patients receiving valproic acid. J Infect Dis. 2007 Mar 15;195(6):833-6. doi: 10.1086/511823. Epub 2007 Jan 30. PMID 17299713
- [Background] Archin NM, Eron JJ, Palmer S, Hartmann-Duff A, Martinson JA, Wiegand A, Bandarenko N, Schmitz JL, Bosch RJ, Landay AL, Coffin JM, Margolis DM. Valproic acid without intensified antiviral therapy has limited impact on persistent HIV infection of resting CD4+ T cells. AIDS. 2008 Jun 19;22(10):1131-5. doi: 10.1097/QAD.0b013e3282fd6df4. PMID 18525258
- [Background] Sagot-Lerolle N, Lamine A, Chaix ML, Boufassa F, Aboulker JP, Costagliola D, Goujard C, Pallier C, Delfraissy JF, Lambotte O; ANRS EP39 study. Prolonged valproic acid treatment does not reduce the size of latent HIV reservoir. AIDS. 2008 Jun 19;22(10):1125-9. doi: 10.1097/QAD.0b013e3282fd6ddc. PMID 18525257
- [Background] Archin NM, Cheema M, Parker D, Wiegand A, Bosch RJ, Coffin JM, Eron J, Cohen M, Margolis DM. Antiretroviral intensification and valproic acid lack sustained effect on residual HIV-1 viremia or resting CD4+ cell infection. PLoS One. 2010 Feb 23;5(2):e9390. doi: 10.1371/journal.pone.0009390. PMID 20186346
- [Background] Archin NM, Espeseth A, Parker D, Cheema M, Hazuda D, Margolis DM. Expression of latent HIV induced by the potent HDAC inhibitor suberoylanilide hydroxamic acid. AIDS Res Hum Retroviruses. 2009 Feb;25(2):207-12. doi: 10.1089/aid.2008.0191. PMID 19239360
- [Background] Contreras X, Schweneker M, Chen CS, McCune JM, Deeks SG, Martin J, Peterlin BM. Suberoylanilide hydroxamic acid reactivates HIV from latently infected cells. J Biol Chem. 2009 Mar 13;284(11):6782-9. doi: 10.1074/jbc.M807898200. Epub 2009 Jan 9. PMID 19136668
- [Background] Chun TW, Carruth L, Finzi D, Shen X, DiGiuseppe JA, Taylor H, Hermankova M, Chadwick K, Margolick J, Quinn TC, Kuo YH, Brookmeyer R, Zeiger MA, Barditch-Crovo P, Siliciano RF. Quantification of latent tissue reservoirs and total body viral load in HIV-1 infection. Nature. 1997 May 8;387(6629):183-8. doi: 10.1038/387183a0. PMID 9144289
- [Background] Archin NM, Bateson R, Tripathy MK, Crooks AM, Yang KH, Dahl NP, Kearney MF, Anderson EM, Coffin JM, Strain MC, Richman DD, Robertson KR, Kashuba AD, Bosch RJ, Hazuda DJ, Kuruc JD, Eron JJ, Margolis DM. HIV-1 expression within resting CD4+ T cells after multiple doses of vorinostat. J Infect Dis. 2014 Sep 1;210(5):728-35. doi: 10.1093/infdis/jiu155. Epub 2014 Mar 11. PMID 24620025
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Kelly WK, O'Connor OA, Krug LM, Chiao JH, Heaney M, Curley T, MacGregore-Cortelli B, Tong W, Secrist JP, Schwartz L, Richardson S, Chu E, Olgac S, Marks PA, Scher H, Richon VM. Phase I study of an oral histone deacetylase inhibitor, suberoylanilide hydroxamic acid, in patients with advanced cancer. J Clin Oncol. 2005 Jun 10;23(17):3923-31. doi: 10.1200/JCO.2005.14.167. Epub 2005 May 16. PMID 15897550
- [Background] Archin NM, Keedy KS, Espeseth A, Dang H, Hazuda DJ, Margolis DM. Expression of latent human immunodeficiency type 1 is induced by novel and selective histone deacetylase inhibitors. AIDS. 2009 Sep 10;23(14):1799-806. doi: 10.1097/QAD.0b013e32832ec1dc. PMID 19590405
- [Background] Shan L, Deng K, Shroff NS, Durand CM, Rabi SA, Yang HC, Zhang H, Margolick JB, Blankson JN, Siliciano RF. Stimulation of HIV-1-specific cytolytic T lymphocytes facilitates elimination of latent viral reservoir after virus reactivation. Immunity. 2012 Mar 23;36(3):491-501. doi: 10.1016/j.immuni.2012.01.014. Epub 2012 Mar 8. PMID 22406268
- [Background] DeBenedette MA, Calderhead DM, Ketteringham H, Gamble AH, Horvatinovich JM, Tcherepanova IY, Nicolette CA, Healey DG. Priming of a novel subset of CD28+ rapidly expanding high-avidity effector memory CTL by post maturation electroporation-CD40L dendritic cells is IL-12 dependent. J Immunol. 2008 Oct 15;181(8):5296-305. doi: 10.4049/jimmunol.181.8.5296. PMID 18832685
- [Background] Calderhead DM, DeBenedette MA, Ketteringham H, Gamble AH, Horvatinovich JM, Tcherepanova IY, Nicolette CA, Healey DG. Cytokine maturation followed by CD40L mRNA electroporation results in a clinically relevant dendritic cell product capable of inducing a potent proinflammatory CTL response. J Immunother. 2008 Oct;31(8):731-41. doi: 10.1097/CJI.0b013e318183db02. PMID 18779746
- [Background] Tcherepanova I, Harris J, Starr A, Cleveland J, Ketteringham H, Calderhead D, Horvatinovich J, Healey D, Nicolette CA. Multiplex RT-PCR amplification of HIV genes to create a completely autologous DC-based immunotherapy for the treatment of HIV infection. PLoS One. 2008 Jan 30;3(1):e1489. doi: 10.1371/journal.pone.0001489. PMID 18231576
- [Background] Addo MM, Yu XG, Rosenberg ES, Walker BD, Altfeld M. Cytotoxic T-lymphocyte (CTL) responses directed against regulatory and accessory proteins in HIV-1 infection. DNA Cell Biol. 2002 Sep;21(9):671-8. doi: 10.1089/104454902760330219. PMID 12396610
- [Background] Van Gulck ER, Ponsaerts P, Heyndrickx L, Vereecken K, Moerman F, De Roo A, Colebunders R, Van den Bosch G, Van Bockstaele DR, Van Tendeloo VF, Allard S, Verrier B, Maranon C, Hoeffel G, Hosmalin A, Berneman ZN, Vanham G. Efficient stimulation of HIV-1-specific T cells using dendritic cells electroporated with mRNA encoding autologous HIV-1 Gag and Env proteins. Blood. 2006 Mar 1;107(5):1818-27. doi: 10.1182/blood-2005-01-0339. Epub 2005 Nov 1. PMID 16263796
- [Background] Altfeld M, Addo MM, Eldridge RL, Yu XG, Thomas S, Khatri A, Strick D, Phillips MN, Cohen GB, Islam SA, Kalams SA, Brander C, Goulder PJ, Rosenberg ES, Walker BD; HIV Study Collaboration. Vpr is preferentially targeted by CTL during HIV-1 infection. J Immunol. 2001 Sep 1;167(5):2743-52. doi: 10.4049/jimmunol.167.5.2743. PMID 11509618
- [Background] Novitsky V, Cao H, Rybak N, Gilbert P, McLane MF, Gaolekwe S, Peter T, Thior I, Ndung'u T, Marlink R, Lee TH, Essex M. Magnitude and frequency of cytotoxic T-lymphocyte responses: identification of immunodominant regions of human immunodeficiency virus type 1 subtype C. J Virol. 2002 Oct;76(20):10155-68. doi: 10.1128/jvi.76.20.10155-10168.2002. PMID 12239290
- [Background] Quaranta MG, Mattioli B, Giordani L, Viora M. The immunoregulatory effects of HIV-1 Nef on dendritic cells and the pathogenesis of AIDS. FASEB J. 2006 Nov;20(13):2198-208. doi: 10.1096/fj.06-6260rev. PMID 17077296
- [Background] Majumder B, Janket ML, Schafer EA, Schaubert K, Huang XL, Kan-Mitchell J, Rinaldo CR Jr, Ayyavoo V. Human immunodeficiency virus type 1 Vpr impairs dendritic cell maturation and T-cell activation: implications for viral immune escape. J Virol. 2005 Jul;79(13):7990-8003. doi: 10.1128/JVI.79.13.7990-8003.2005. PMID 15956545
- [Background] Tcherepanova I, Starr A, Lackford B, Adams MD, Routy JP, Boulassel MR, Calderhead D, Healey D, Nicolette C. The immunosuppressive properties of the HIV Vpr protein are linked to a single highly conserved residue, R90. PLoS One. 2009 Jun 10;4(6):e5853. doi: 10.1371/journal.pone.0005853. PMID 19516896
- [Background] Routy JP, Boulassel MR, Yassine-Diab B, Nicolette C, Healey D, Jain R, Landry C, Yegorov O, Tcherepanova I, Monesmith T, Finke L, Sekaly RP. Immunologic activity and safety of autologous HIV RNA-electroporated dendritic cells in HIV-1 infected patients receiving antiretroviral therapy. Clin Immunol. 2010 Feb;134(2):140-7. doi: 10.1016/j.clim.2009.09.009. Epub 2009 Nov 4. PMID 19889582
- [Background] Jones RB, O'Connor R, Mueller S, Foley M, Szeto GL, Karel D, Lichterfeld M, Kovacs C, Ostrowski MA, Trocha A, Irvine DJ, Walker BD. Histone deacetylase inhibitors impair the elimination of HIV-infected cells by cytotoxic T-lymphocytes. PLoS Pathog. 2014 Aug 14;10(8):e1004287. doi: 10.1371/journal.ppat.1004287. eCollection 2014 Aug. PMID 25122219
- [Background] Rasmussen TA, Schmeltz Sogaard O, Brinkmann C, Wightman F, Lewin SR, Melchjorsen J, Dinarello C, Ostergaard L, Tolstrup M. Comparison of HDAC inhibitors in clinical development: effect on HIV production in latently infected cells and T-cell activation. Hum Vaccin Immunother. 2013 May;9(5):993-1001. doi: 10.4161/hv.23800. Epub 2013 Jan 31. PMID 23370291
- [Background] Elliott JH, Wightman F, Solomon A, Ghneim K, Ahlers J, Cameron MJ, Smith MZ, Spelman T, McMahon J, Velayudham P, Brown G, Roney J, Watson J, Prince MH, Hoy JF, Chomont N, Fromentin R, Procopio FA, Zeidan J, Palmer S, Odevall L, Johnstone RW, Martin BP, Sinclair E, Deeks SG, Hazuda DJ, Cameron PU, Sekaly RP, Lewin SR. Activation of HIV transcription with short-course vorinostat in HIV-infected patients on suppressive antiretroviral therapy. PLoS Pathog. 2014 Nov 13;10(10):e1004473. doi: 10.1371/journal.ppat.1004473. eCollection 2014 Oct. PMID 25393648
- [Background] Sogaard O, Graversen ME, Leth S, Brinkmann C, Kjaer AS, Olesen R, et al. The HDAC inhibitor romidepsin is safe and effectively reverses HIV-1 latency in vivo as measured by standard clinical assays. In: 20th International AIDS Conference. Melbourne, Australia; 2014.
- [Background] Wei DG, Chiang V, Fyne E, Balakrishnan M, Barnes T, Graupe M, Hesselgesser J, Irrinki A, Murry JP, Stepan G, Stray KM, Tsai A, Yu H, Spindler J, Kearney M, Spina CA, McMahon D, Lalezari J, Sloan D, Mellors J, Geleziunas R, Cihlar T. Histone deacetylase inhibitor romidepsin induces HIV expression in CD4 T cells from patients on suppressive antiretroviral therapy at concentrations achieved by clinical dosing. PLoS Pathog. 2014 Apr 10;10(4):e1004071. doi: 10.1371/journal.ppat.1004071. eCollection 2014 Apr. PMID 24722454
- [Background] Cillo AR, Krishnan S, McMahon DK, Mitsuyasu RT, Para MF, Mellors JW. Impact of chemotherapy for HIV-1 related lymphoma on residual viremia and cellular HIV-1 DNA in patients on suppressive antiretroviral therapy. PLoS One. 2014 Mar 17;9(3):e92118. doi: 10.1371/journal.pone.0092118. eCollection 2014. PMID 24638072
- [Background] Bullen CK, Laird GM, Durand CM, Siliciano JD, Siliciano RF. New ex vivo approaches distinguish effective and ineffective single agents for reversing HIV-1 latency in vivo. Nat Med. 2014 Apr;20(4):425-9. doi: 10.1038/nm.3489. Epub 2014 Mar 23. PMID 24658076
- [Background] Debenedette M, Tcherepanova I, Gamble AH, Horatinovich J, Harris J, Routy JP, et al. Immune function and viral load post AGS-004 administration to chronic HIV subjects undergoing STI. In: 2014 Conference on Retroviruses and Opportunistic Infections. Boston, MA; 2014.
- [Background] Marks P, Rifkind RA, Richon VM, Breslow R, Miller T, Kelly WK. Histone deacetylases and cancer: causes and therapies. Nat Rev Cancer. 2001 Dec;1(3):194-202. doi: 10.1038/35106079. PMID 11902574
- [Background] Richon VM, Emiliani S, Verdin E, Webb Y, Breslow R, Rifkind RA, Marks PA. A class of hybrid polar inducers of transformed cell differentiation inhibits histone deacetylases. Proc Natl Acad Sci U S A. 1998 Mar 17;95(6):3003-7. doi: 10.1073/pnas.95.6.3003. PMID 9501205
- [Background] Secrist JP, Zhou X, Richon VM. HDAC inhibitors for the treatment of cancer. Curr Opin Investig Drugs. 2003 Dec;4(12):1422-7. PMID 14763127
- [Background] Munster PN, Troso-Sandoval T, Rosen N, Rifkind R, Marks PA, Richon VM. The histone deacetylase inhibitor suberoylanilide hydroxamic acid induces differentiation of human breast cancer cells. Cancer Res. 2001 Dec 1;61(23):8492-7. PMID 11731433
- [Background] He LZ, Tolentino T, Grayson P, Zhong S, Warrell RP Jr, Rifkind RA, Marks PA, Richon VM, Pandolfi PP. Histone deacetylase inhibitors induce remission in transgenic models of therapy-resistant acute promyelocytic leukemia. J Clin Invest. 2001 Nov;108(9):1321-30. doi: 10.1172/JCI11537. PMID 11696577
- [Background] Ruefli AA, Ausserlechner MJ, Bernhard D, Sutton VR, Tainton KM, Kofler R, Smyth MJ, Johnstone RW. The histone deacetylase inhibitor and chemotherapeutic agent suberoylanilide hydroxamic acid (SAHA) induces a cell-death pathway characterized by cleavage of Bid and production of reactive oxygen species. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10833-8. doi: 10.1073/pnas.191208598. Epub 2001 Sep 4. PMID 11535817
- [Background] Huang L, Pardee AB. Suberoylanilide hydroxamic acid as a potential therapeutic agent for human breast cancer treatment. Mol Med. 2000 Oct;6(10):849-66. PMID 11126200
- [Background] Butler LM, Agus DB, Scher HI, Higgins B, Rose A, Cordon-Cardo C, Thaler HT, Rifkind RA, Marks PA, Richon VM. Suberoylanilide hydroxamic acid, an inhibitor of histone deacetylase, suppresses the growth of prostate cancer cells in vitro and in vivo. Cancer Res. 2000 Sep 15;60(18):5165-70. PMID 11016644
- [Background] Vrana JA, Decker RH, Johnson CR, Wang Z, Jarvis WD, Richon VM, Ehinger M, Fisher PB, Grant S. Induction of apoptosis in U937 human leukemia cells by suberoylanilide hydroxamic acid (SAHA) proceeds through pathways that are regulated by Bcl-2/Bcl-XL, c-Jun, and p21CIP1, but independent of p53. Oncogene. 1999 Nov 25;18(50):7016-25. doi: 10.1038/sj.onc.1203176. PMID 10597302
- [Background] Mitsiades N, Mitsiades CS, Richardson PG, McMullan C, Poulaki V, Fanourakis G, Schlossman R, Chauhan D, Munshi NC, Hideshima T, Richon VM, Marks PA, Anderson KC. Molecular sequelae of histone deacetylase inhibition in human malignant B cells. Blood. 2003 May 15;101(10):4055-62. doi: 10.1182/blood-2002-11-3514. Epub 2003 Jan 16. PMID 12531799
- [Background] Lindemann RK, Gabrielli B, Johnstone RW. Histone-deacetylase inhibitors for the treatment of cancer. Cell Cycle. 2004 Jun;3(6):779-88. Epub 2004 Jun 14. PMID 15153801
- [Background] Warrener R, Beamish H, Burgess A, Waterhouse NJ, Giles N, Fairlie D, Gabrielli B. Tumor cell-selective cytotoxicity by targeting cell cycle checkpoints. FASEB J. 2003 Aug;17(11):1550-2. doi: 10.1096/fj.02-1003fje. Epub 2003 Jun 3. PMID 12824307
- [Background] Glaser KB, Staver MJ, Waring JF, Stender J, Ulrich RG, Davidsen SK. Gene expression profiling of multiple histone deacetylase (HDAC) inhibitors: defining a common gene set produced by HDAC inhibition in T24 and MDA carcinoma cell lines. Mol Cancer Ther. 2003 Feb;2(2):151-63. PMID 12589032
- [Background] Bali P, Pranpat M, Bradner J, Balasis M, Fiskus W, Guo F, Rocha K, Kumaraswamy S, Boyapalle S, Atadja P, Seto E, Bhalla K. Inhibition of histone deacetylase 6 acetylates and disrupts the chaperone function of heat shock protein 90: a novel basis for antileukemia activity of histone deacetylase inhibitors. J Biol Chem. 2005 Jul 22;280(29):26729-34. doi: 10.1074/jbc.C500186200. Epub 2005 Jun 2. PMID 15937340
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Archin NM, Crooks AM, Bateson R, Cope AB, Dahl NP, Eron J, et al. Measuring HIV Latency Over Time: Reservoir Stability and Assessing Interventions. In: Conference on Retroviruses and Opportunistic Infections. Boston, MA; 2014.
- [Background] Gandhi RT, Zheng L, Bosch RJ, Chan ES, Margolis DM, Read S, Kallungal B, Palmer S, Medvik K, Lederman MM, Alatrakchi N, Jacobson JM, Wiegand A, Kearney M, Coffin JM, Mellors JW, Eron JJ; AIDS Clinical Trials Group A5244 team. The effect of raltegravir intensification on low-level residual viremia in HIV-infected patients on antiretroviral therapy: a randomized controlled trial. PLoS Med. 2010 Aug 10;7(8):e1000321. doi: 10.1371/journal.pmed.1000321. PMID 20711481